CLINICAL TRIAL: NCT05722938
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center, Phase III Trial to Assess the Efficacy and Safety of Trimodulin (BT588) in Adult Hospitalized Subjects With Severe Community-acquired Pneumonia (sCAP)
Brief Title: Efficacy and Safety of Trimodulin (BT588) in Subjects With Severe Community-acquired Pneumonia (sCAP)
Acronym: ESsCAPE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 996
Record Dates: First submitted 2023-01-11; First posted 2023-02-10 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Community-acquired Pneumonia
Keywords: Severe Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — trimodulin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized on a 1:1 basis to receive trimodulin or placebo, stratified by center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All bottles will be indistinguishable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trimodulin (Experimental): Trimodulin (human IgM, IgA, IgG solution) for intravenous (IV) administration.
  Interventions: Drug: Trimodulin
- Placebo (Placebo Comparator): Human albumin 1%
  Interventions: Drug: Placebo (human albumin 1%)

INTERVENTIONS:
Drug: Trimodulin — IMP will be administered via IV infusion on 5 consecutive days
  Other Names: BT588
  Arms: Trimodulin
Drug: Placebo (human albumin 1%) — IMP will be administered via IV infusion on 5 consecutive days
  Arms: Placebo

SUMMARY:
The main objective of the trial is to assess the efficacy and safety of trimodulin as adjunctive treatment to standard of care (SoC) compared to placebo plus SoC in adult hospitalized subjects with sCAP on invasive mechanical ventilation (IMV).

Other objectives are to determine detailed pharmacokinetic (PK) properties of trimodulin in a PK substudy and to determine its pharmacodynamic (PD) properties.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multi-center, multi-national, phase III trial, to assess the efficacy and safety of trimodulin compared to placebo treatment, as adjunctive treatment to SoC in adult hospitalized subjects with sCAP receiving IMV.

Subjects will be randomized on a 1:1 basis to receive trimodulin or placebo, stratified by center. Investigational medicinal product (IMP) treatments will be blinded.

Subject will be administered IMP once daily on 5 consecutive days (day 1 through day 5) adjunctive to SoC. The subsequent follow-up phase comprises maximally 23 days (day 6 through day 28) followed by an end-of-follow-up visit/telephone call on day 29 [+3]. For subjects still in the hospital (trial site) after day 29, an extended follow-up is conducted until discharge or until day 90. For all subjects alive on day 29, a closing visit/telephone call on day 91 [+10] will be done.

ELIGIBILITY:
Main Inclusion Criteria:

1. Written informed consent.
2. Hospitalized, adult (≥ 18 years of age) subject.
3. Signs of inflammation based on C-reactive protein threshold level.
4. Diagnosis of active community-acquired pneumonia (CAP) before hospital-admission or within 48 hours after admission.
5. Radiological (or other imaging technology) evidence consistent with active pneumonia.
6. Acute respiratory failure requiring IMV.

Main Exclusion Criteria:

1. For an incapacitated subject: any indication that the subject's presumed will would be against inclusion in the trial.
2. Pregnant or lactating women.
3. Subjects of childbearing potential not willing to use reliable contraceptive measures during the trial and for 15 weeks after the last IMP treatment.
4. Subjects on ECMO or predicted to be on ECMO at start of IMP treatment.
5. Suspected hospital-acquired pneumonia (HAP) including ventilator-associated pneumonia (VAP).
6. Subjects discharged from hospital within the previous 14 days.
7. Defined neutrophil counts within 24 hours prior to start of IMP treatment.
8. Defined platelet counts within 24 hours prior to start of IMP treatment.
9. Defined hemoglobin within 24 hours prior to start of IMP treatment.
10. Pre-existing hemolytic disease.
11. Pre-existing thrombosis or other thromboembolic events (TEEs) within 3 months before start of IMP treatment. Subjects particularly at risk for TEEs caused by other reasons than the current sCAP.
12. Subject on dialysis or with severe renal impairment within 24 hours prior to start of IMP treatment.
13. Subject with end-stage renal disease (ESRD) or known primary focal segmental glomerulosclerosis (FSGS).
14. Pre-existing severe lung diseases concomitant to current sCAP (e.g., subjects with chronic obstructive pulmonary disease [COPD] Gold Stage III or IV, severe interstitial lung disease [incl. idiopathic pulmonary fibrosis], cystic fibrosis, active tuberculosis, chronically infected bronchiectasis, or active lung cancer).
15. Pre-existing decompensated heart failure.
16. Pre-existing severe hepatic cirrhosis (Child Pugh score ≥ 10 points), or severe hepatic impairment (Child Pugh score ≥ 10 points), or hepatocellular carcinoma.
17. Known intolerance to proteins of human origin or known allergic reactions to components of trimodulin / placebo.
18. Selective immunoglobulin A (IgA) deficiency with known antibodies to IgA.
19. Life expectancy of less than 90 days, according to the investigator's clinical judgment, because of medical conditions related neither to sCAP nor to sCAP-associated septic conditions.
20. Morbid obesity with high body mass index (BMI) ≥ 40 kg/m2, or malnutrition with low BMI < 16 kg/m2.
21. Treatment with polyvalent immunoglobulin preparations during the last 21 days before start of IMP treatment.
22. Known treatment with predefined medications, during the last 2 days before start of IMP treatment.
23. Treatment with any type of interferon during the last 21 days before start of IMP treatment
24. Subject with previous organ or hematopoietic stem cell transplantation receiving ongoing treatment with immunosuppressants (exception: corticosteroids) at start of IMP treatment.
25. Participation in another interventional clinical trial (using medications and/or procedures not according to SoC of the trial site) within 30 days before start of IMP treatment or previous IMP treatment in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality rate | Between days 1-29
  Percentage of subjects that died until day 29 regardless of cause of death

SECONDARY OUTCOMES:
90-day all-cause mortality rate | Between days 1-91
  Percentage of subjects that died until day 91 regardless of cause of death
28-day all-cause mortality rate plus day 6-29 deterioration rate | 1. Between days 1-29; 2. Between days 6-29
  1. Percentage of subjects that died until day 29
  2. Percentage of subjects with at least one deterioration event between day 6 and day 29
Deterioration rate (day 6-29) | Between days 6-29
  Percentage of subjects with at least one deterioration event between day 6 and day 29
28-day all-cause mortality rate plus day 1-29 deterioration rate | 1.+2. Between days 1-29
  1. Percentage of subjects that died until day 29
  2. Percentage of subjects with at least one deterioration event between day 1 and day 29
Deterioration rate (day 1-29) | Between days 1-29
  Percentage of subjects with at least one deterioration event between day 1 and day 29
Change in Sequential Organ Failure Assessment (SOFA) score from baseline to days 3, 5, 7, 14, 21, 29 and discharge | Between baseline and Days 3, 5, 7, 14, 21, 29 and discharge
  Change in Sequential Organ Failure Assessment (SOFA)
Proportion of subjects with clinical cure of pneumonia on days 7, 14, 21, 29 and discharge | On days 7, 14, 21, 29 or on the day of discharge
  Percentage of subjects with clinical cure of pneumonia
Days of invasive mechanical ventilation (IMV) until day 29 | Until day 29
  Days of invasive mechanical ventilation (IMV) until day 29
Ventilator-free days (VFD) until day 29 | Until day 29
  Ventilator-free days (VFD)
Days with oxygen supply until day 29 | Until day 29
  Days with oxygen supply
Proportion of subjects with oxygen supply on days 7, 14, 21, 29 and discharge | On days 7, 14, 21, 29 or on the day of discharge
  Percentage of subjects with oxygen supply
Proportion of subjects with PaO2/FiO2 ratio < 100, 100 to < 200, 200 to < 300 or ≥ 300 on days 7, 14, 21, and 29 | On days 7, 14, 21, 29
  Percentage of subjects with PaO2/FiO2 ratio < 100, 100 to < 200, 200 to < 300 or ≥ 300
Vasopressor-free days until day 29 | Until day 29
  Vasopressor-free days until day 29
Days in intensive care unit (ICU) until day 29 | Until day 29
  Days in intensive care unit (ICU) until day 29
Time to discharge from ICU | Until day 91
  Time to discharge from ICU
Proportion of subjects in ICU on days 7, 14, 21 and 29 | On days 7, 14, 21, 29
  Percentage of subjects in ICU
Days of hospitalization until day 29 | Until day 29
  Days of hospitalization
Time to discharge from hospital | Until day 91
  Time to discharge from hospital
Proportion of subjects in hospital on days 7, 14, 21 and 29 | On days 7, 14, 21, 29
  Percentage of subjects in hospital
28-day readmission rate | Day 29
  Percentage of subjects readmitted to the hospital
Rate of unscheduled return(s) to the emergency department or primary physician between day 29 and day 91 | Between Days 29 - 91
  Percentage of subjects returning to the emergency department or primary physician
Time to return to normal activities until day 91 | Until day 91
  Time to return to normal activities
Health status based on Clinical Frailty Scale (CFS) on day 91 | Between Days 29 - 91
  Change in Health status from Baseline assessment based on Clinical Frailty Scale (score 1 very fit to score 9 terminally ill)
Quality of life based on Nottingham Health Profile (NHP) on days 29 and 91 | Day 29 and day 91
  Change in Quality of life based on Nottingham Health Profile (NHP)
Adverse events (AEs), treatment-emergent AEs (TEAEs), AEs of special interest (AESIs), infusional TEAEs, TEAEs that led to permanent withdrawal of IMP and/or discontinuation of trial | Until day 29
  Number, severity, causality, outcome, and seriousness of all AEs and TEAEs, AESIs, infusional TEAEs, TEAEs that led to permanent withdrawal of IMP, and TEAEs that led to discontinuation of the trial
Infusion-related TEAEs | Until day 29
  Number of all infusion-related TEAEs
Serious adverse events (SAEs) | Until day 29
  Number, severity, causality, and outcome of all SAEs
Dose modifications | Day 1-5
  Dose modifications (including reductions and changes in infusion rate)
Change over time in electrocardiogram (ECG) parameters | Days -1, 1, 3, 5 and once between days 8-13
  ECG output (diagram including QT-interval and QTcF) showing abnormal, clinically relevant findings will be reported as adverse event
Number and changes in observed Adverse Events in vital signs over time | Days -1, 1-3, 5, 7, 14, 21, 29
  Clinically significant changes in values of vital signs (including systolic and diastolic blood pressure, arterial oxygen saturation, heart rate, respiratory rate and body temperature) are rated as adverse events. The number of adverse events and changes in numbers of the adverse events over time will be reported
Number and changes in observed Adverse Events in clinical laboratory parameters over time | Days -1, 1-5, 7, 14, 21, 29
  Clinically significant changes in clinical laboratory values (including chemistry, hematology and coagulation) are rated as adverse events. The number of adverse events and changes in numbers of the adverse events over time will be reported

OTHER OUTCOMES:
Serum concentration of immunoglobulins | Day 1, 5, 14
  Changes of serum concentration of IgM, IgA, and IgG from baseline, during and after treatment
Pharmacokinetic assessment of immunoglobulins | Day 1, 2, 3, 4, 5, 6, 7, 9, 14, 21, 29
  Assessment of changes in serum concentrations (g/L) of IgM, IgA, and IgG before, during and after treatment
Pharmacodynamic assessment of disease related serum proteins | Day 1, 2, 3, 4, 5, 7, 14, 21, 29
  Assessment of relative changes in serum concentrations from baseline, during and after treatment of factors and markers of coagulation (e.g. % change in D-dimer), markers of inflammation (e.g. % change in CRP), complement factors (e.g. % change in C3, C4), specific antibody titers against sCAP-related pathogens (e.g. % change in Streptococcus pneumoniae antibody titers)

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Ferrer Roca, Dr., Principal Investigator — Hospital Vall d'Hebron
Locations (146):
- United States (19):
  - Pulmonary Associates of Mobile, P.C., Mobile, Alabama
  - University of California San Francisco-Fresno, Fresno, California
  - UC Davis Health, Sacramento, California
  - Augusta University, Augusta, Georgia
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Missouri Clinical Research Center, Columbia, Missouri
  - Hannibal Clinic, Hannibal, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - St. Michael's Medical Center, Newark, New Jersey
  - Buffalo VA Medical Center, Buffalo, New York
  - Lenox Hill Hospital, New York, New York
  - Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medical City Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Argentina (12):
  - Sanatorio Parque S.A. Privado, San Vicente, Córdoba Province
  - CEMIC, Ciudad Autonoma de Buenos Aire
  - Sanatorio de la Trinidad Mitre, Ciudad Autonoma de Buenos Aire
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire
  - Hospital General de Agudos Dr. Ignacio Pirovano, Ciudad Autonoma de Buenos Aire
  - Clinica Adventista Belgrano, Ciudad Autonoma de Buenos Aire
  - Clinica Chutro, Córdoba
  - Hospital San Roque, Córdoba
  - Sanatorio Privado de la Canada - Cordoba, Córdoba
  - Centro Medico IPAM, Rosario
  - Estudios Clinicos de los Arroyos, San Nicolás
  - Sanatorio de la Canada, Villa María
- Australia (6):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Footscray Hospital, Footscray
  - Austin Health, Heidelberg
  - Sunshine Hospital, Saint Albans
- Austria (2):
  - KABEG-Klinikum Klagenfurt, Klagenfurt
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (12):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - AZ Sint-Jan, Bruges
  - Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital (UZA), Edegem
  - ZOL, Genk
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - C. H. R. de la Citadelle, Liège
  - CHU Charleroi Hôpital Civil Marie Curie, Lodelinsart
  - Clinique Saint-Pierre, Ottignies
  - AZ Delta VZW, Roeselare
- Brazil (11):
  - UPECLIN - Unidade de Pesquisa Clínica, Botucatu
  - HMCP - Hospital e Maternidade Celso Pierro - PUC-Campinas, Campinas
  - Hospital do Rocio, Campo Largo
  - Universidade de Caxias do Sul, IPCEM - Instituto de Pesquisa Clínica para Estudos Multicêntricos, Caxias do Sul
  - Hospital de Clínicas de Passo Fundo, Passo Fundo
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - CIP - Centro Integrado de Pesquisa, São José do Rio Preto
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Universidade Municipal de Sao Caetano do Sul (USCS), São Paulo
- Czechia (4):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Oblastni nemocnice Kolin a.s., Kolín
  - Hospital Kyjov, Kyjov
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- France (20):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Hôpital Louis Mourier, Colombes
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CHRU Lille - Hôpital Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier de Melun, Melun
  - CHU Nice-Hopital de l' Archet, Nice
  - CHU Nice Hopital Pasteur 2, Nice
  - Hôpital Bichat - Claude Bernard, Paris
  - Groupe Hospitalier Diaconesses - Hopital De La Croix Saint Simon, Paris
  - Hôpital Tenon, Paris
  - Hôpital Cochin, Paris
  - CHU Reims - Hôpital Robert Debré, Reims
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg
  - Hôpital Sainte Musse, Toulon
  - CHU Tours - Hôpital Bretonneau, Tours
  - Hôpital Nord Franche-Comté, Trévenans
- Germany (5):
  - Charité Universitätsmedizin Berlin - Campus Charité Mitte, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Hungary (6):
  - Bugat Pal Korhaz, Gyöngyös
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Aneszteziologiai es Intenziv Terapias Intezet, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Ireland (4):
  - St James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - St Vincents University Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- New Zealand (2):
  - Middlemore Hospital, Otahuhu
  - Capital, Coast and Hutt Valley District - Wellington Regional Hospital, Wellington
- Philippines (8):
  - Baguio General Hospital and Medical Center, Baguio City
  - Dr. Jose N. Rodriguez Memorial Hospital, Caloocan
  - Davao Doctors Hospital, Davao City
  - Southern Philippines Medical Center, Davao City
  - St.Paul's Hospital, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Philippine General Hospital, Manila
  - Lung Center of the Philippines, Quezon City
- Romania (3):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic Judetean de Urgenta "Pius Brinzeu", Timișoara
- South Africa (7):
  - Johese Clinical Research, Centurion, Gauteng
  - Emmed Clinical Research, Pretoria, Gauteng
  - Into Research, Pretoria, Gauteng
  - Worthwhile Clinical Trials, Johannesburg
  - RYEXO Clinical Research Zuid Afrikaans Hospital, Pretoria
  - RYEXO Clinical Research, Pretoria
  - Dr JM Engelbrecht Trial Site, Somerset West
- Spain (14):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Universitari Mutua de Terrassa, Terrassa
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - Queen Elizabeth University Campus, Glasgow
  - Royal Surrey County Hospital, Guildford
  - St Thomas' Hospital, London
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No